CLINICAL TRIAL: NCT01748370
Title: A Randomized, Double-blind, Placebo Controlled Trial to Evaluate the Effects of Vitamin D Supplementation on Androgen Levels in Hypogonadal Men
Brief Title: Vitamin D Treatment and Hypogonadism in Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lerchbaum Elisabeth, MD, Clinical Professor, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VitDTesto1.0; 14846 (Other Grant/Funding Number: ÖNB Jubiläumsfond)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Hypogonadism
Keywords: vitamin D; hypogonadism; testosterone; intervention
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D hypogonadal (Experimental): Vitamin D supplementation in hypogonadal men
  Interventions: Drug: Vitamin D supplementation in hypogonadal men
- Vitamin D eugonadal (Experimental): Vitamin D supplementation in eugonadal men
  Interventions: Drug: Vitamin D supplementation in eugonadal men
- Placebo hypogonadal (Placebo Comparator): Vitamin D supplementation in hypogonadal men
  Interventions: Drug: Placebo hypogonadal
- Placebo eugonadal (Placebo Comparator): Vitamin D supplementation in eugonadal men
  Interventions: Drug: Placebo eugonadal

INTERVENTIONS:
Drug: Vitamin D supplementation in hypogonadal men
  Other Names: A11CC05 Colecalciferol
  Arms: Vitamin D hypogonadal
Drug: Vitamin D supplementation in eugonadal men
  Other Names: A11CC05 Colecalciferol
  Arms: Vitamin D eugonadal
Drug: Placebo hypogonadal
  Arms: Placebo hypogonadal
Drug: Placebo eugonadal
  Arms: Placebo eugonadal

SUMMARY:
Low total testosterone (TT) is present in about 30% of men aged >60 years and in up to 7% of younger men. Male hypogonadism is associated with metabolic and cardiovascular diseases as well as with increased mortality. There is evidence showing a relationship of TT with vitamin D in men. We aim at evaluating the effect of vitamin D supplementation on TT and metabolic parameters in hypogonadal men. We will study the effects of 20,000 IU vitamin D weekly in a 12 wk randomized, double-blind, placebo-controlled trial in 100 men with TT <3.0 ng/ml and 25-hydroxyvitamin D (25(OH)D) <30 ng/ml (patients) as well as in 100 men with TT ≥3.0 ng/ml and 25(OH)D <30 ng/ml (controls). Vitamin D supplementation might be a safe therapeutic approach improving TT levels as well as metabolic parameters in hypogonadal men. Further the effects of vitamin D on androgens will be evaluated in eugonadal men.

ELIGIBILITY:
Hypogonadal men:

Inclusion Criteria:

* TT levels below 3.0 ng/ml (measured at the baseline visit and confirmed at study visit 1)
* 25(OH)D levels below 30 ng/ml (measured at the baseline visit)
* Male, age of ≥ 18 and <70 years
* Written informed consent before entered into study

Exclusion Criteria:

* - Hypercalcemia defined as a serum calcium > 2,7 mmol/L
* Oral or transdermal testosterone supplementation in the last 2 months before entering the study
* IM testosterone supplementation 6 months before entering the study
* Regular intake of vitamin D supplements before study entry
* Men with chronic diseases (such as diabetes mellitus, thyroid disease, endocrine disturbances in need of treatment (except hypogonadism), or diseases known to interfere with vitamin D intake or very sensitive to vitamin D intake (such as inflammatory disease with granuloma: sarcoidoses, tuberculosis, Mb Wegener, vasculitis, inflammatory bowel disease
* Intake of medication influencing metabolic or endocrine parameters (insulin sensitizers, insulin, glucocorticoids,…) in the last 3 months before study entry
* PSA >4 ng/ml (or >3 ng/ml in men at high risk for prostate cancer) (see state of the art)
* Palpable prostate nodule or induration
* Hematocrit >50%
* Untreated severe obstructive sleep apnea
* Severe lower urinary tract symptoms
* Uncontrolled or poorly controlled heart failure
* A history of prostate cancer, breast cancer, orchidectomy, chromosomal disorders (e.g. Klinefelter Syndrome)

Eugonadal men:

Inclusion Criteria:

* TT levels ≥3.0 ng/ml (measured at the baseline visit and confirmed at study visit 1)
* 25(OH)D levels below 30 ng/ml (measured at the baseline visit)
* Male, age of ≥ 18 and <70 years
* Written informed consent before entered into study

Exclusion Criteria:

* Hypercalcemia defined as a serum calcium > 2,7 mmol/L
* Oral or transdermal testosterone supplementation in the last 2 months before entering the study
* IM testosterone supplementation 6 months before entering the study
* Regular intake of vitamin D supplements before study entry
* Men with chronic diseases (such as diabetes mellitus, endocrine disturbances in need of treatment (except hypogonadism), or diseases known to interfere with vitamin D intake or very sensitive to vitamin D intake (such as inflammatory disease with granuloma: sarcoidoses, tuberculosis, Mb Wegener, vasculitis, inflammatory bowel disease
* Intake of medication influencing metabolic or endocrine parameters (insulin sensitizers, insulin, glucocorticoids,…) in the last 3 months before study entry
* PSA >4 ng/ml (or >3 ng/ml in men at high risk for prostate cancer) (see state of the art)
* Palpable prostate nodule or induration
* Hematocrit >50%
* Untreated severe obstructive sleep apnea
* Severe lower urinary tract symptoms
* Uncontrolled or poorly controlled heart failure
* A history of prostate cancer, breast cancer, orchidectomy, chromosomal disorders (e.g. Klinefelter)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
Total testosterone (TT) | Change from baseline in TT at 12 weeks

SECONDARY OUTCOMES:
Free testosterone (FT) | Change from baseline in FT after 12 weeks
Insulin resistance assessed by homeostatic model assessment-insulin resistance (HOMA-IR) | Change from baseline in HOMA-IR at 12 weeks
Lipid levels (total cholesterol) | Change from baseline in total cholesterol at 12 weeks
Metabolic response during an oral glucose tolerance test (oGTT) as defined by AUCgluc | Change from Baseline in AUCgluc at 12 weeks
Metabolic response during an oral glucose tolerance test (oGTT) as defined by AUCins | Change from Baseline in AUCins at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Lerchbaum, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department of Internal Medicine, Division of Endocrinology and Metabolism, Graz, Austria

REFERENCES:
- [Derived] Lerchbaum E, Pilz S, Trummer C, Schwetz V, Pachernegg O, Heijboer AC, Obermayer-Pietsch B. Vitamin D and Testosterone in Healthy Men: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2017 Nov 1;102(11):4292-4302. doi: 10.1210/jc.2017-01428. PMID 28938446